CLINICAL TRIAL: NCT04131829
Title: Brain Network Changes Accompanying and Predicting Responses to Pharmacotherapy in OCD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000023688; 1R01MH116038-01A1 (NIH); 1K24MH121571-01 (NIH)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fluoxetine

STUDY DESIGN:
Intervention Model Description: 80 OCD patients and 40 healthy participants matched on demographics will be recruited and asked to complete Structural (sMRI) and Functional (fMRI) Magnetic Resonance Imaging. Patients with OCD will be randomized to immediate monotherapy or 6-week placebo-delayed monotherapy, with fluoxetine.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy Controls (No Intervention): The healthy control group will be an age matched sample of unmedicated healthy adults who will be recruited and imaged once at baseline and the data compared with that of OCD subjects at baseline.
- OCD Group (Experimental): The OCD group will comprise of unmedicated individuals with clinically significant OCD symptoms. OCD Subjects will be randomized, double-blind, to receive immediate or delayed (by 6 weeks as a placebo lead-in) pharmacotherapy.
  Interventions: Drug: Fluoxetine - immediate treatment; Drug: Fluoxetine - delayed treatment

INTERVENTIONS:
Drug: Fluoxetine - immediate treatment — Following the Baseline assessment, OCD subjects will be randomized to receive either immediate fluoxetine monotherapy or delayed fluoxetine, after a 6-week placebo lead-in.
  Other Names: fluoxetine, prozac
  Arms: OCD Group
Drug: Fluoxetine - delayed treatment — Following the Baseline assessment, OCD subjects will be randomized to receive either immediate fluoxetine monotherapy or delayed fluoxetine, after a 6-week placebo lead-in.
  Other Names: fluoxetine, prozac
  Arms: OCD Group

SUMMARY:
The proposed randomized, double-blind research study will use functional magnetic resonance neuroimaging using state-of-the-art HCP acquisition protocols and analytic pipelines, to identify predictors and correlates of response to an accepted first-line pharmacological treatment for obsessive-compulsive disorder.

DETAILED DESCRIPTION:
The proposed study intends to recruit 2 groups:

1. Matched healthy control participants will be imaged with one fMRI at baseline as a no-treatment comparison group; and
2. a randomized, double-blind group of unmedicated OCD participants who will be assigned to begin either immediate or placebo-delayed treatment, and who will be imaged with fMRIs at baseline and over the course of treatment with a selective serotonin reuptake inhibitor (SSRI), fluoxetine.

Hypothesis-driven analyses and exploratory analyses will be performed in parallel.

This study will address the following Specific Aims:

1. Identification of neural dysconnectivity associated with OCD symptomatology.
2. Characterizing neural markers of clinical response to SSRI pharmacotherapy.
3. Mapping neural predictors of clinical response to pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for all groups will include: (i) Adults, Men and women will be included, in a 1:1 ratio; and efforts will be made to recruit racial and ethnic subgroups. Groups will be further matched on age, handedness; and later, in analysis, on educational status and smoking history.

(ii) signed informed consent, approved by the Yale Human Investigations Committee; and (iii) ability and willingness to participate in all study procedures, including clinical assessments and fMRI scans.

* Additional inclusion criteria:
* OCD Participants:

  (i) a DSM diagnosis of OCD, established as detailed above; (ii) a baseline Y-BOCS of ≥16; (iii) no current psychoactive medication, with the exception of the occasional use of a PRN medication for sleep; (iv) treatment seeking, and clinically appropriate for fluoxetine pharmacotherapy; (v) for women of childbearing potential, not pregnant or intending to become pregnant, and willing to use reliable birth control over the course of the study, either prescribed contraceptive (oral contraceptive, injectable, or implant) or one barrier method (e.g. diaphragm with spermicide, intrauterine device, cervical cap). Women of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy tests at the study baseline and on each scan day appointment prior to the MRI scan.
* Healthy Control Participants:

  (i) no current DSM diagnosis (by clinician interview confirmed by SCID or MINI); (ii) no documented or clinically suspected family history in a first- or second- degree relative of OCD, Tourette syndrome, hoarding disorder, body dysmorphic disorder, or a compulsive grooming disorder.

Exclusion Criteria:

* Exclusion criteria for all groups will include:

  (i) any unstable medical, psychiatric, or neurological condition (including active or otherwise problematic suicidality) that may necessitate urgent treatment; (ii) any substance use disorder within the past 6 months; (iii) use of psychotropic medications within the past 8 weeks, with the exception of occasional use of a sleep aid or analgesic; (iv) use of an as-needed sleep aid or prescription analgesic within 3 days of the scan; (v) any history of a primary psychotic disorder or of mania; (vi) any evidence of substance use on urine toxicology testing; (vii) any major neurological disease or history of major head trauma, including concussion with extended loss of consciousness; (viii) pregnancy; (ix) any metal in the body or other contraindication to MRI scanning; (x) severe claustrophobia, back pain, or other condition that may make an extended MR scan difficult or lead to excessive movement during the scan.
* Additional exclusion criteria:
* OCD Participants:

  (i) past allergy or adverse reaction to fluoxetine or another SSRI, or other clinical contraindication to fluoxetine pharmacotherapy; (ii) documented nonresponse to a past trial of fluoxetine of appropriate dose (≥40 mg/dy) and duration (≥12 weeks).

(iii) Patients taking Coumadin or Monoamine oxidase inhibitors (MAOIs) will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Obsessive-compulsive severity change | 18 weeks
  Yale-Brown Obsessive-Compulsive Scale (Y-BOCS);72,73 -This is a checklist and Clinician administered - 10 item severity scale, from none to extreme. Total severity score range is 0 to 40. This will be presented as % improvement in Y-BOCS as a continuous measure of treatment response, rather than an artificially dichotomized measure of 'response', in all analyses. This the primary outcome measure of change across the study treatment and scans.

SECONDARY OUTCOMES:
Tic severity change | 18 weeks
  Yale Global Tic Severity Scale (YGTSS) will be used to measure Tic severity. It is a clinician administered instrument with a score from 0 to 25- 25 being the most severe.
Beck Depression Inventory-II | 18 weeks
  Beck Depression Inventory-II (BDI-II);82 21 items to assess intensity of depression.
Anxiety | 18 weeks
  Beck Anxiety Inventory (BAI);83 21 item self report on a 4 point Likert scale - 0 (not at all) to 3 (severely).
Obsessive-compulsive concerns | 18 weeks
  Dimensional Obsessive-Compulsive Scale (DOCS);84 20 questions, asks about 4 categories of obsessive-compulsive concerns (each consists of 5 items scored on a Likert scale of 0-no symptoms to 4 - extreme symptoms) over the previous month.
Magical ideation | 18 weeks
  Magical Ideation Scale (MIS);86 30 item true / false scale, assessing erroneous beliefs based on magical thinking.
Sensory phenomena | 18 weeks
  University of São Paulo Sensory Phenomena Scale (USP-SPS);87
"Not Just Right" experiences and sensations in OCD | 18 weeks
  Not Just Right Experiences Questionnaire Revised (INC).88 19 Questions: Rate 10 NJR Experiences; Choose most recent one; Identify how long ago it occurred; then complete 7 dimensional ratings of that NJRE: frequency, intensity, immediate distress, delayed distress, rumination, urge to respond, and responsibility to do something about the NJRE, from 1 (absence) to 7 (extreme level /or within the past day).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pittenger, MD, PhD, Principal Investigator — Professor of Psychiatry; Director, Yale OCD Research Clinic
Locations (1):
- Yale OCD Research Clinic - CMHC/CNRU, 34 Park ST, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No